CLINICAL TRIAL: NCT05536011
Title: WAKIX® (Pitolisant) Pregnancy Registry: An Observational Study of the Safety of Pitolisant Exposure in Pregnant Women and Their Offspring
Brief Title: WAKIX® (Pitolisant) Pregnancy Registry
Status: Recruiting | Type: Observational
Sponsor: Harmony Biosciences Management, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: HBS-101-CL-008
Record Dates: First submitted 2022-09-07; First posted 2022-09-10 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Pregnancy Related; Narcolepsy
MeSH Terms: conditions — Narcolepsy | interventions — pitolisant; Modafinil; Sodium Oxybate; solriamfetol; Methylphenidate; Amphetamines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 21 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (5):
- Pitolisant-exposed participants with narcolepsy: Pregnant women with a diagnosis of narcolepsy who are exposed to pitolisant at any time during pregnancy
  Interventions: Drug: Pitolisant
- Unexposed participants with narcolepsy: Pregnant women with a diagnosis of narcolepsy who are not exposed to pitolisant or a comparator product at any time during pregnancy
- Comparator-exposed participants with narcolepsy: Pregnant women with a diagnosis of narcolepsy who are not exposed to pitolisant at any time during pregnancy but who are exposed to comparator products at any time during pregnancy
  Interventions: Drug: Comparator Products
- Pitolisant-exposed participants without narcolepsy: Pregnant women without a diagnosis of narcolepsy who are exposed to pitolisant at any time during pregnancy
  Interventions: Drug: Pitolisant
- Comparator-exposed participants without narcolepsy: Pregnant women without a diagnosis of narcolepsy who are not exposed to pitolisant at any time during pregnancy but who are exposed to a comparator product at any time during pregnancy
  Interventions: Drug: Comparator Products

INTERVENTIONS:
Drug: Pitolisant — Exposure to at least one dose of pitolisant at any time during pregnancy
  Other Names: Wakix
  Groups: Pitolisant-exposed participants with narcolepsy; Pitolisant-exposed participants without narcolepsy
Drug: Comparator Products — Exposure to at least one dose of a comparator product at any time during pregnancy
  Other Names: Modafinil/armodafinil; Sodium oxybate; Oxybate mixed salts; Solriamfetol; Methylphenidate; Amphetamines
  Groups: Comparator-exposed participants with narcolepsy; Comparator-exposed participants without narcolepsy

SUMMARY:
The WAKIX (pitolisant) Pregnancy Registry is a US-based, prospective, observational cohort study designed to evaluate the association between pitolisant exposure during pregnancy and subsequent maternal, fetal, and infant outcomes.

DETAILED DESCRIPTION:
The WAKIX (pitolisant) Pregnancy Registry is a US-based, prospective, observational cohort study designed to evaluate the association between pitolisant exposure during pregnancy and subsequent maternal, fetal, and infant outcomes. Participation in the registry is voluntary and participants can withdraw their consent to participate at any time. Data will be collected from enrolled pregnant women and the healthcare providers (HCPs) involved in their care or the care of their infants, if applicable. The registry is strictly observational; the schedule of office visits and all treatment regimens will be determined by HCPs. Only data that are routinely documented in patients' medical records during the course of usual care will be collected. No additional laboratory tests or HCP assessments will be required as part of this registry. The design of this pregnancy registry follows current FDA guidance for designing and implementing pregnancy exposure registries.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant woman of any age
* Consent to participate
* Authorization for her HCP(s) to provide data to the registry
* For participants with a diagnosis of narcolepsy: exposure to at least one dose of pitolisant or one dose of a comparator product, or, unexposed to pitolisant or comparator products at any time during pregnancy (i.e., any pregnant woman with a diagnosis of narcolepsy)
* For participants without a diagnosis of narcolepsy: exposure to at least one dose of pitolisant or one dose of a comparator product at any time during pregnancy

Exclusion Criterion:

• Occurrence of pregnancy outcome prior to first contact with the Registry Coordination Center (RCC) (i.e., retrospectively enrolled)

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The narcolepsy study population will include three cohorts (cohort 1, 2 and 3) of pregnant women with a diagnosis of narcolepsy:
  * Cohort 1, exposed to pitolisant at any time during pregnancy
  * Cohort 2, unexposed to pitolisant or any comparator product at any time during pregnancy
  * Cohort 3, unexposed to pitolisant but exposed to a comparator product at any time during pregnancy
  The non-narcolepsy study population will include two cohorts (cohorts 4 and 5) of pregnant women without a diagnosis of narcolepsy:
  * Cohort 4, exposed to pitolisant at any time during pregnancy
  * Cohort 5, unexposed to pitolisant but exposed to a comparator product at any time during pregnancy
Sampling Method: Non-Probability Sample
Enrollment: 1329 (Estimated)
Dates: Start 2021-08-24 (Actual); Primary Completion 2030-06-30 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
Major congenital malformation | Enrollment through the infant's first year of life
  An abnormality of body structure or function that is present at birth, is of prenatal origin (i.e., birth defect), has significant medical, social, or cosmetic consequences for the affected individual, and typically requires medical intervention.

SECONDARY OUTCOMES:
Minor congenital malformation | Enrollment through the infant's first year of life
  An anomaly or abnormality of body structure that is present at birth, is of prenatal origin (i.e., birth defect), poses no significant health problem in the neonatal period, and tends to have limited social or cosmetic consequences for the affected individual.
Pre-eclampsia | Enrollment through pregnancy outcome
  High blood pressure and signs of liver or kidney damage occurring at >20 gestational weeks.
Eclampsia | Enrollment through pregnancy outcome
  Seizures or coma in a pregnant woman with pre-eclampsia.
Spontaneous abortion | Enrollment through pregnancy outcome
  An involuntary fetal loss or the expulsion of the products of conception occurring at <20 gestational weeks.
Stillbirth | Enrollment through pregnancy outcome
  As defined by the American College of Obstetricians and Gynecologists (ACOG), an involuntary fetal loss occurring at ≥20 gestational weeks or, if gestational age is unknown, a fetus weighing ≥350 g.
Elective termination | Enrollment through pregnancy outcome
  A voluntary fetal loss or interruption of pregnancy, including pregnancy termination that occurs electively, to preserve maternal health or due to fetal abnormalities.
Preterm birth | Enrollment through the infant's first year of life
  A live birth occurring at <37 gestational weeks.
Small for gestational age | Enrollment through the infant's first year of life
  Weight, length, or head circumference at birth in <10th percentile for sex and gestational age using standard growth charts for full and preterm live born infants.
Postnatal growth deficiency | Enrollment through the infant's first year of life
  Weight, length, or head circumference in <10th percentile for sex and chronological age using standard growth charts
Infant development deficiency | Enrollment through the infant's first year of life
  Failure to achieve the developmental milestones for chronological age, as defined by the Centers for Disease Control and Prevention (CDC).

CONTACTS AND LOCATIONS:
Locations (1):
- Evidera (PPD), Morrisville, North Carolina, United States